CLINICAL TRIAL: NCT03871101
Title: Evaluation of Dental Anxiety in Patients Undergoing Second Stage Surgery With Er,Cr:YSGG Laser Treatment: Randomized Clinical Trial
Brief Title: Evaluation of Dental Anxiety in Second-Stage Implant Surgery With Er,Cr:YSGG Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Erkan Feslihan, Principal investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24112017-02
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Dental Anxiety
Keywords: Dental Anxiety; STAI; Er,Cr:YSGG; oral surgery
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Scalpel (Active Comparator): Soft tissue incision with scalpel in second- stage implant surgery.
  Interventions: Procedure: Scalpel
- Erbium laser (Experimental): Soft tissue incision with 2780 nm Er,Cr:YSGG laser, at implant recovery settings (2.00 W power, 100 Hz H mode, 10% water and 10% air) in second-stage implant surgery.
  Interventions: Device: 2780 nm Er,Cr:YSGG Laser

INTERVENTIONS:
Procedure: Scalpel — Exposure of the cover screw of osseointegrated dental implants embedded under oral mucosa by performing the soft tissue incision with scalpel for placing the healing abutment.
  Arms: Scalpel
Device: 2780 nm Er,Cr:YSGG Laser — Exposure of the cover screw of osseointegrated dental implants embedded under oral mucosa by performing the soft tissue incision with erbium laser for placing the healing abutment.
  Arms: Erbium laser

SUMMARY:
Implants embedded under the oral mucosa were exposed with scalpel (Group 1) or laser surgery (Group 2). Before the operation the patients were asked to fill the State-Trait Anxiety Inventory (STAI) and Dental Anxiety Scale (DAS) while resting in the waiting room.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing second-stage implant surgery

Exclusion Criteria:

* Patients without sufficient keratinized gingiva
* Bone overlap on closure screw
* Implants that can not be localized due to gingiva thickness,

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Dental anxiety | 20 minutes before the operation
  Before the operation the patients were asked to fill the State-Trait Anxiety Inventory (STAI) questionary.Patients' answers to each question were scored between 1-4 points. A total of 20-37 anxiety scores were assessed as minimum level of anxiety or none, 38-44 points as moderate and 45-80 as high.
Dental Anxiety | 20 minutes before the operation
  Before the operation the patients were asked to fill the Dental Anxiety Scale (DAS). Patients' answers to questions were scored between 1-4 points. The total score of the questions in the questionnaire ranged from 4 to 20, and 4-11 points were interpreted as low level dental anxiety, 12-14 points as moderate and more than 14 points as high.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet C Talmac, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University Faculty of Dentistry, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Candido MC, Andreatini R, Zielak JC, de Souza JF, Losso EM. Assessment of anxiety in patients who undergo surgical procedures for tooth implants: a prospective study. Oral Maxillofac Surg. 2015 Sep;19(3):253-8. doi: 10.1007/s10006-014-0480-3. Epub 2015 Jan 10. PMID 25572978
- [Background] Kazancioglu HO, Dahhan AS, Acar AH. How could multimedia information about dental implant surgery effects patients' anxiety level? Med Oral Patol Oral Cir Bucal. 2017 Jan 1;22(1):e102-e107. doi: 10.4317/medoral.21254. PMID 27918733

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03871101/Prot_SAP_000.pdf